CLINICAL TRIAL: NCT02829567
Title: Effectiveness of Motivational Interviewing in Improving Oral Hygiene in Orthodontic Patients
Brief Title: Motivational Interviewing in Orthodontic Patients
Acronym: MIOrtho
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Barcelona (Other)
Responsible Party: Principal Investigator, Maria Montserrat Rigau Gay, DDS, University of Barcelona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MI01
Record Dates: First submitted 2016-06-26; First posted 2016-07-12 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-04

CONDITIONS: Oral Hygiene
MeSH Terms: interventions — Motivational Interviewing

ARMS (2):
- Oral hygiene counseling and motivational interviewing (Experimental): This group will receive a session of oral hygiene counseling and a single session of motivational interviewing to increase the readiness of change.
  Interventions: Behavioral: Motivational interviewing
- Oral hygiene counseling (No Intervention)

INTERVENTIONS:
Behavioral: Motivational interviewing
  Arms: Oral hygiene counseling and motivational interviewing

SUMMARY:
The purpose of this study is to determine whether motivational interviewing is effective in improving oral hygiene in orthodontic patients wearing fixed appliances.

ELIGIBILITY:
Inclusion Criteria:

* Orthodontic patients wearing fixed appliances, within the first six months of treatment
* Eruption completed (except for the third molars) or late mixed dentition.
* Caucasian

Exclusion Criteria:

* Pregnancy
* Periodontal disease
* Systemic illness
* Medical treatment

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 130 (Actual)
Dates: Start 2016-01; Primary Completion 2017-12 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Assess change in oral hygiene using plaque index Löe & Silness | Baseline, 1 month and 6 months
  Plaque index Löe & Silness (Time: baseline, 1 month and 6 months)

SECONDARY OUTCOMES:
Assess change in oral hygiene using gingival index Löe & Silness | Baseline, 1 month and 6 months
  Gingival index Löe & Silness ( Time: baseline, 1 month and 6 months)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Montserrat Rigau Gay, DDS, Principal Investigator — University of Barcelona
Locations (1):
- Hospital Odontològic Universitat de Barcelona, L'Hospitalet de Llobregat, Barcelona, Spain

REFERENCES:
- [Background] Martins RK, McNeil DW. Review of Motivational Interviewing in promoting health behaviors. Clin Psychol Rev. 2009 Jun;29(4):283-93. doi: 10.1016/j.cpr.2009.02.001. Epub 2009 Feb 23. PMID 19328605
- [Derived] Rigau-Gay MM, Claver-Garrido E, Benet M, Lusilla-Palacios P, Ustrell-Torrent JM. Effectiveness of motivational interviewing to improve oral hygiene in orthodontic patients: A randomized controlled trial. J Health Psychol. 2020 Nov-Dec;25(13-14):2362-2373. doi: 10.1177/1359105318793719. Epub 2018 Sep 10. PMID 30198774